CLINICAL TRIAL: NCT05384431
Title: Can We Achieve 'high-quality' Weight Loss Through Supplementation and Exercise? the TRIM MUSCLE Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Exerkine Corporation (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 43396
Record Dates: First submitted 2022-05-10; First posted 2022-05-20 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Exercise; Supplementation; Aerobic training; Resistance training; Insulin sensitivity; Sex differences; Inflammation; Oxidative stress; Weight management; Antioxidants; Protein
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Insulin Resistance; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, parallel group design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All Exerkine and University of Waterloo research staff will be blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Muscle5 and TRIM7 (Active Comparator): MUSCLE5 and TRIM7 natural health product supplementation
  Name of natural health product (brand name, generic) - MUSCLE 5, chocolate Is this a market-approved natural health product (per Health Canada)? - Yes Dose - 1 scoop Ingredients (per dose) - Whey protein isolate (24g), milk protein isolate (16g), Creatine (3g), Calcium (450mg), Vitamin D (1000 IU) Frequency of administration - Once/day Duration (e.g., six weeks) - 12 weeks Route of administration - Oral
  Name of natural health product (brand name, generic) - TRIM7 Is this a market-approved natural health product (as per Health Canada)? Yes Dose - 3 capsules Ingredients (per dose) - Alpha lipoic acid (200mg), CoEnzyme Q10 (100mg), beet root extract (250mg), green coffee bean extract (250mg), green tea extract (250mg), forskolin (25mg), Vitamin E (22 mg AT) Frequency of administration - Twice/day Duration (e.g., six weeks) - 12 weeks Route of administration - Oral
  Interventions: Dietary Supplement: Muscle5 and TRIM7; Other: Mixed exercise
- Placebo (Placebo Comparator): Placebo collagen and microcrystalline cellulose intake
  Placebo Control 1 (Counter to MUSCLE5) Dose - 1 scoop Ingredients (per dose) - Collagen (40g) Frequency of administration - once/day Duration - 12 weeks Route of administration - Oral
  Placebo Control 2 (Counter to TRIM7) Dose - 3 capsules Ingredients (per dose) - Microcrystalline cellulose (400 mg) Frequency of administration - twice/day Duration - 12 weeks Route of administration - Oral
  Interventions: Other: Mixed exercise

INTERVENTIONS:
Dietary Supplement: Muscle5 and TRIM7 — Intake of MUSCLE 5 and TRIM 7 supplements on a daily basis for 12 weeks
  Arms: Muscle5 and TRIM7
Other: Mixed exercise — Mixed exercise (aerobic and resistance) three days per week for 12 weeks

SUMMARY:
The purpose of this study is to determine whether the combination of two dietary supplements: MUSCLE 5, which contains protein, creatine and vitamin D and TRIM 7, which contains beet extract, caffeine, coenzyme Q10, alpha lipoic acid, forskolin extract, green coffee bean extract, green tea and vitamin E, plus exercise can induce greater 'high-quality' weight loss than exercise alone in overweight and obese men and women. First, the investigators will examine whether the addition of these two supplements to a mixed exercise regime (e.g., aerobic and resistance training) induces greater improvements in typical training adaptations (aerobic capacity, upper & lower body muscle strength, lean mass, ASM, fat mass, % body fat, and lean mass/fat mass). Secondly, the investigators will assess improvements in pro- and anti-inflammatory factors, insulin sensitivity, and blood lipids. Third, the investigators will determine effects on perceived stress, sleep quality, hair & nail growth, and health-related quality of life. Overweight men and women will be randomized to either exercise alone or exercise plus supplement for 12 weeks. Training will include mixed exercise (aerobic and resistance) three days per week and supplements will be taken on a daily basis. Before and after the 12-week training period the investigators will assess A) Body weight, BMI, DXA outcomes (total lean mass, total body fat, % body fat, ASM, and lean mass/fat mass), waist circumference, VO2max, and upper/lower body maximal strength, B) Circulatory inflammatory factors, antioxidants, blood lipids, and oral glucose tolerance/insulin sensitivity (OGTT), C) Perceived stress, sleep quality, hair & nail growth, and health-related quality of life and D) Overall Health Index. Benefits of the study to participants may include weight loss and improved health (irrespective of weight loss). Benefits of the study to the scientific community include improved understanding of how high-quality protein- and antioxidant-containing supplements, combined with mixed exercise, affect weight loss and overall health in men and women. Thus, the investigators will be comparing men and women to determine if the response to supplementation and exercise is similar or different between the sexes.

DETAILED DESCRIPTION:
The purpose of the proposed study is to determine if the addition of two supplements (TRIM 7 and MUSCLE 5) to an exercise regime can induce more favorable effects on body weight, BMI, body composition (lean mass, fat mass, % body fat, ASM, and lean mass/fat mass), upper & lower body strength, aerobic fitness (VO2max), insulin sensitivity (OGTT), blood lipids (cholesterol and triglycerides), antioxidant capacity (total reducing capacity of plasma), inflammation (TNFα, IL6, CRP, IL- 10) and overall health in overweight men and women.

Primary objective/research question*:

-Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater 'high-quality' weight loss?

Co-primary objectives/research questions*:

* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater loss of bodyweight?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater improvement in body mass index (BMI)?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater improvement in waist-to-hip ratio?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater loss of fat mass?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program maintain or improve lean mass?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program maintain or improve lean mass/fat mass ratio (e.g., body composition index)?

Secondary objectives/research questions:

* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater improvements in muscle strength and aerobic capacity?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater improvements in insulin sensitivity?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater reductions in inflammation and greater increases in antioxidant status?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater improvements in sleep quality, perceived stress, health-related quality of life and the overall health index?
* Can the addition of TRIM 7 and MUSCLE 5 to an exercise program induce greater improvements in hair & nail growth?

Hypotheses:

* The addition of TRIM 7 and MUSCLE 5 will induce greater 'high-quality' weight loss than exercise alone as evidenced by A) greater loss of fat mass, B) greater gain (or maintenance) of lean mass, C) greater improvement in lean mass/fat mass ratio (e.g., body composition index) D) greater loss of bodyweight E) greater reduction in waist-to-hip ratio and/or F) greater improvement in BMI.
* The addition of TRIM 7 and MUSCLE 5 will induce greater improvements in muscle strength and aerobic fitness than exercise alone as evidenced by a greater improvement in 1RM and VO2peak than exercise alone.
* The addition of TRIM 7 and MUSCLE 5 will induce greater improvements in insulin sensitivity (HOMA-IR, glycemic control during an OGTT, Matsuda Index) than exercise alone.
* The addition of TRIM 7 and MUSCLE 5 will induce a greater reduction in inflammation (TNFα, IL6, CRP, IL- 10) and induce a greater improvement in antioxidant status (GSH:GSSG, CuZn SOD, MnSOD, catalase, total reducing capacity of plasma) than exercise alone.
* The addition of TRIM 7 and MUSCLE 5 will induce greater improvements in sleep quality, perceived stress, health-related quality of life, and an overall health index than exercise alone.
* The addition of TRIM 7 and MUSCLE 5 will induce greater improvements in hair & nail growth than exercise alone.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 45 years
* BMI > 25 kg/m2
* low physical activity level < 150 min/week (< ACSM and CSEP recommendations)
* have had two doses of the COVID-19 vaccine

Exclusion Criteria:

* renal disease (creatinine > 140)
* liver disease (i.e. diagnosed NAFLD, NASH, cirrhosis, previous liver transplant)
* GI disorders (i.e. Colitis, Crohns)
* cardiovascular disease (recent myocardial infarction (< 6 months), hypertension requiring more than 2 medications, congestive heart failure requiring more than one medication for control, unstable arrhythmia, angina previous stroke with residual hemiparesis)
* severe osteoarthritis
* significant weight loss in the 3-month period prior to the study (10% of total body weight)
* muscular dystrophy
* severe peripheral neuropathy
* severe osteoporosis
* uncontrolled hypertension (>140/90 mmHg)
* orthopedic problems
* type I or II diabetes
* respiratory conditions (i.e. chronic pulmonary obstructive disorder), chronic obstructive pulmonary disease (FVC or FEV1 < 70% of age predicted mean value), and asthma requiring more than two medications
* individuals with prior bariatric surgery
* women who have ammenorrhea, dysregulated menstrual cycle, are peri-menopausal, menopausal, pregnant, looking to become pregnant, or nursing
* medications, including anti-inflammatory medications, more than one glucose lowering medication, insulin, platelet inhibitors, anti-coagulant medications, or Simvastatin (zocor), beta-blockers, or weight loss medications (Orlistat, Saxenda Contrave) or any other medications known to affect protein metabolism (i.e.corticosteroids).
* inability to take part in the exercise program
* vegan
* smoking
* history of glaucoma or
* overactive bladder syndrome
* consumption of more than 10 drinks/week or 2 drinks/d for women and 15 drinks/week or 3 drinks/d for men.
* history of allergy, sensitivity or strong dislike towards any component of the study products (supplements)
* have undergone a barium swallow or an infusion of a contrast agent in the past 3 weeks
* have an implantable electronic device
* inability to perform exercise as determined by the Get Active Questionnaire (GAQ)
* inability to consent
* participants on volitional dietary supplements will be considered on a case-by-case basis, but they will be asked to refrain from intake for at least 2 weeks prior to partaking in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Bodyweight change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  scale
BMI change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  Body mass index (weight/height squared)
Fat mass change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  body composition by DEXA
Lean mass change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  body composition by DEXA
Lean mass/fat mass (body composition index) change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  body composition by DEXA
Percent body fat change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  body composition by DEXA
Waist-to-hip ratio change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  measure tape

SECONDARY OUTCOMES:
VO2max change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  Maximal aerobic capacity test (gas exchange and indirect calorimetry measured using a metabolic cart and incremental cycle ergometry)
Lower body strength change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  1-repetition and 5-repetition maximal strength
Upper body strength change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  1-repitition maximal strength and 5-repeitition maximal strength
Appendicular lean mass change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  body composition by DEXA
Insulin sensitivity change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  Oral glucose tolerance test (OGTT)
Blood lipids change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  cholesterol (LDL, HDL, and total cholesterol) and triglycerides
Inflammation CRP change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  pro-inflammatory circulatory factor (ng/mL) by Luminex Performance Assay
Inflammation TNF-alpha change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  pro inflammatory circulatory factor (pg/ml) by Luminex Performance Assay
Inflammation IL-1 change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  pro inflammatory circulatory factor (pg/ml) by Luminex Performance Assay
Inflammation IL-10 change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  anti-inflammatory circulatory factors (pg/mL) by Luminex Performance Assay
Inflammation IL-6 change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  pro-inflammatory circulatory factor (pg/mL) by Luminex Performance Assay
Antioxidant capacity change | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  TEAC (trolox equivalent antioxidant assay)

OTHER OUTCOMES:
Perceived stress change (Perceived Stress Scale) | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  Perceived Stress Scale (PSS-10; 0 = lowest stress, 40 = highest stress)
Sleep quality change (Bergen Insomnia Scale) | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  Bergen Insomnia Scale (0 = lowest insomnia, 42 = highest insomnia)
Health-related quality of life (SF 36) | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  36 Item Short Form Survey (SF 36; 0 = maximal disability, 100 = no disability)
Male hair growth & quality (Merk & Co, 1996) | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  5 item survey (Merk & Co; 38 = maximal score (highest quality), 5 = lowest score (lowest quality))
Female hair growth & quality (WHGQ) | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  4 item survey (WHGQ; 28 = maximal score (highest quality), 4 = lowest score (lowest quality))
Nail health | baseline 0 weeks ("pre study") to 12 weeks ("post study")
  5 item survey (25 = maximal score, 5 = lowest score)
Nail growth change | baseline 0 weeks ("pre study"), 6 weeks ("midway"), and 12 weeks ("post study")
  Ten-day nail growth will be measured by a digital caliper (Mitotoyu 500) three times during the course of the study (baseline, midway, and post).

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Devries-Aboud, PhD, Principal Investigator — Kinesiology and Health Sciences, University of Waterloo
Locations (1):
- Michaela Devries-Aboud, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There are no plans of making the clinical trial data at the individual level available to researchers who were not part of the original study team